CLINICAL TRIAL: NCT01659762
Title: A Phase I Study Evaluating Safety and Tolerability of Autologous Bone Marrow Derived Mesenchymal Stromal (MSC) Cells in Adults With Moderate to Severe Crohn's Disease.
Brief Title: A Phase I Study Evaluating Autologous Bone Marrow Derived Mesenchymal Stromal for Crohn's Disease.
Acronym: EPIC/MSC/IBD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Atlanta Clinical and Translational Science Institute (Other)
Responsible Party: Principal Investigator, Jacques Galipeau, MD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00051454; EPIC001 (Other: Other)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Crohn's Disease
Keywords: inflammatory bowel disease; Crohn's disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous mesenchymal stromal cells (Experimental)
  Interventions: Biological: autologous mesenchymal stromal cell

INTERVENTIONS:
Biological: autologous mesenchymal stromal cell

SUMMARY:
In this Phase I trial the investigators intend to show safety and tolerability of autologous MSC, expanded using a non-xenogeneic, human component platelet lysate expansion media. Fresh, non cryopreserved, autologous MSCs will delivered intravenously as a single bolus dose in a dose escalation phase I study. The investigators intend to test whether the product is clinically safe in adults (18-65 years old) with CD and to determine maximal deliverable dose. Secondary endpoint will monitor effectiveness using CDAI as an endpoint.

DETAILED DESCRIPTION:
EPIC MSC/IBD is made up of autologous marrow-derived mesenchymal stromal cells ex vivo expanded numerically for approximately 14 days using pooled human Platelet Lysate (phPL), harvested on the day of infusion, washed and suspended at a concentration of 4 million cells/ml in Plasmalyte A with 0.5% human serum albumin. This is a phase I dose-escalation, open label, non-randomized, non-placebo controlled, single group assignment study to evaluate the safety and tolerability of a single intravenous infusion of EPIC MSC2011-001. EPIC EPIC MSC/IBD will be infused intravenously and will be administered at one of three dose levels: (Tier 1) 2 million cells/kg patient body weight; (Tier 2) 5 million cells/kg, and (Tier 3) 10 million cells/kg. This Phase I clinical trial will enroll 16-20 subjects with moderate to severe Crohn's. The duration of this study for each patient is 12 weeks. The investigators anticipate that this study will be completed within 2 years of commencement.

Primary objective: To describe and compare the safety and tolerability of a single infusion of fresh autologous bone marrow derived Mesenchymal stromal cells infused to patients with moderate to severe Crohn's disease.

Secondary objective: Efficacy of autologous bone marrow derived Mesenchymal stromal cells infusion to patients with moderate to severe Crohn's disease as assessed through disease activity index, and quality of life index.

Safety variables:Adverse events (AEs),Laboratory parameters (hematology, biochemistry, urinalysis), Vital signs.

ELIGIBILITY:
Inclusion Criteria

* Men and women 18-65 years of age.
* Patient must have had CD for at least 3 months from the time of initial diagnosis. The diagnosis of CD must have been confirmed by endoscopic and histological evidence.
* Patients must have active Crohn's disease as defined by a Crohns Disease Activity Index (CDAI) score between >220 at screening and baseline.
* Patients should have no need for immediate surgery (i.e. due to obstruction, strictures, active abscess or perforations ).
* Subjects must be refractory (defined as lack of response for at least 3 months) to immunomodulators (including 6-mercaptopurine and azathioprine and methotrexate) or anti-TNF therapy at present or some point in the course of their disease. Lack of response is defined by failure to reduce the CDAI score by at least 70 points.
* The following medications will be allowed: mesalamine and prednisone (stable dose for at least 2 weeks prior to enrollment).
* Subjects on anti TNF therapy will require a minimum of 4 weeks washout period prior to screening.
* Subjects on non-steroidal analgesics require a minimum of 2 weeks washout period prior to screening
* If female and of child-bearing age, patient must be non-pregnant, non-breastfeeding, and use adequate contraception;
* Patient is willing to participate in the study and has signed the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 12 months
  Monitoring for adverse events at time of MSC infusion and in 12 months following

SECONDARY OUTCOMES:
Crohn's disease activity Index (CDAI) | 12 months
  CDAI score before and after intervention will be monitored over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Subra Kugathasan, MD, Principal Investigator — Emory University; Tanvi Dhere, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Dhere T, Copland I, Garcia M, Chiang KY, Chinnadurai R, Prasad M, Galipeau J, Kugathasan S. The safety of autologous and metabolically fit bone marrow mesenchymal stromal cells in medically refractory Crohn's disease - a phase 1 trial with three doses. Aliment Pharmacol Ther. 2016 Sep;44(5):471-81. doi: 10.1111/apt.13717. Epub 2016 Jul 7. PMID 27385373